CLINICAL TRIAL: NCT03822637
Title: The Effect of NAC on Lung Function and CT Mucus Score
Acronym: ENACT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to COVID restrictions and funding challenges. The study was then simplified and redesigned as the TEAM study (NCT06152653).
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-26680
Record Dates: First submitted 2018-12-14; First posted 2019-01-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — N-monoacetylcystine; Albuterol; Acetylcysteine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 20% n-acetylcystine (NAC) (Experimental): NAC (trade name: Mucomyst) is manufactured by American Regent. The active drug studied here is 20% NAC coadministered with albuterol and delivered via nebulizer three times per day for fourteen days.
  Interventions: Drug: n-acetylcystine + albuterol
- 0.9% saline (Placebo Comparator): Normal saline will be coadministered with albuterol as the placebo agent via a nebulizer three times per day for fourteen days.
  Interventions: Drug: 0.9% saline + albuterol

INTERVENTIONS:
Drug: n-acetylcystine + albuterol — NAC is a mucolytic drug and Albuterol is a bronchodilator.
  Other Names: Mucomyst; NAC; n-acetylcystine
  Arms: 20% n-acetylcystine (NAC)
Drug: 0.9% saline + albuterol — Normal saline is a placebo agent and Albuterol is a bronchodilator.
  Other Names: Normal saline
  Arms: 0.9% saline

SUMMARY:
This study evaluates 20% n-acetylcysteine (NAC) in the treatment of moderate-to-severe asthma that is complicated by mucus in the airway, as determined by CT imaging. The study is a crossover design, which means that half the study participants will get 20% NAC in the first 14-day treatment period and placebo in the next 14-day treatment period; and the other half will get placebo in the first 14-day treatment period and 20% NAC in the next 14-day treatment period.

DETAILED DESCRIPTION:
N-acetylcystine (NAC) is a mucolytic medication, meaning that it breaks apart mucus. Investigators know that mucus is a factor in severe asthma attacks. However, mucus may be a factor in chronic severe asthma as well. This role has been hard to prove because of difficulty in showing that mucus occludes the lumen in chronic severe disease. Using a novel approach of scoring mucus occlusion, investigators have used CT imaging to uncover that a majority of people with severe asthma have at least one lung segment with a mucus plug and 27% have more than four lung segments with mucus plugs.

Historically, studies of mucolytics, like NAC, have not shown benefit in other obstructive lung diseases, like Chronic Obstructive Pulmonary Disease (COPD). However, utilizing CT mucus scores as a biomarker, investigators believe that mucolytic treatment may prove useful for those with significant mucus impaction.

This is a randomized, double-blind, placebo-controlled phase 4 study of 20% NAC in patients with asthma who also have evidence of mucus in their lungs as determined by CT imaging. Investigators hypothesize that by treating asthmatics, chosen based on the presence of mucus in the airways, with a mucolytic like NAC, will result in an improvement of lung function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 80 years of age at Visit 1
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
3. Able to perform reproducible spirometry according to American Thoracic Society (ATS) criteria
4. Physiological evidence of airflow obstruction (FEV1 bronchodilator reversibility of ≥ 12% or hyperreactivity to methacholine reflected by a methacholine provocative concentration that results in a 20% fall in FEV1(PC20) ≤ 16 mg/mL)
5. Clinical history of asthma per patient report or medical record
6. Pre-bronchodilator FEV1 > 35% predicted
7. Post-bronchodilator FEV1 > 40% but < 90% predicted
8. Asthma requiring treatment with inhaled corticosteroids (ICS) for 3 months or greater
9. CT mucus score ≥ 5
10. Ability to tolerate study drug reflected by a post-treatment FEV1 ≥ 80% of pre- treatment, pre-bronchodilator FEV1

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
3. Smoking of tobacco or other recreational inhalants in last year and/or >10 pack-year smoking history
4. Adherence to study drug ≤ 70% after first treatment period
5. Current participation in an investigational drug trial
6. Other chronic pulmonary disorders, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways
7. Unwillingness to follow study procedures
8. History of allergy or intolerance to study drug
9. Any other criteria that places the subject at unnecessary risk according to the judgment of the Principal Investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 | Through study completion, an average of 9 weeks
  The primary outcome is the % change in FEV1 from the start to the end of each two-week treatment period (either placebo or 20% NAC).

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, M.D, M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hays SR, Fahy JV. The role of mucus in fatal asthma. Am J Med. 2003 Jul;115(1):68-9. doi: 10.1016/s0002-9343(03)00260-2. No abstract available. PMID 12867239
- [Background] DUNNILL MS. The pathology of asthma, with special reference to changes in the bronchial mucosa. J Clin Pathol. 1960 Jan;13(1):27-33. doi: 10.1136/jcp.13.1.27. PMID 13818688